CLINICAL TRIAL: NCT06281314
Title: VESPA 2.0 - Virtual Environment for a Superior Neuropsychiatry Second Generation
Brief Title: The Efficacy of VESPA 2.0 for Cognitive Rehabilitation in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesco Corallo, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VESPA 2.0
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Neurodegenerative Diseases; Cognitive Decline; Parkinson Disease Dementia; Alzheimer Disease; Multiple Sclerosis
MeSH Terms: conditions — Neurodegenerative Diseases; Cognitive Dysfunction; Alzheimer Disease; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson'disease group (Experimental): Rehabilitation takes place with individual one-hour sessions per day. The stimulation intervention is organized on 4 different themes (chosen from orientation, memory, praxis, language, executive functions, attention, problem-solving, and functional activities) for 15' each.
  Interventions: Device: Vespa software
- Multiple Sclerosis group (Experimental): Rehabilitation takes place with individual one-hour sessions per day. The stimulation intervention is organized on 4 different themes (chosen from orientation, memory, praxis, language, executive functions, attention, problem-solving, and functional activities) for 15' each.
  Interventions: Device: Vespa software
- Alzheimer group (Experimental): Rehabilitation takes place with individual one-hour sessions per day. The stimulation intervention is organized on 4 different themes (chosen from orientation, memory, praxis, language, executive functions, attention, problem-solving, and functional activities) for 15' each.
  Interventions: Device: Vespa software

INTERVENTIONS:
Device: Vespa software — The Vespa2.0 project refers to the production of tasks useful for neuropsychological rehabilitation, aimed at subjects suffering from Alzheimer's Dementia, Parkinson's and Multiple Sclerosis. It is a neuropsychological rehabilitation project using Virtual Reality (VR).

SUMMARY:
VESPA 2.0 is based on an integrative and ecological approach used for the treatment of cognitive dysfunction in patients with MCI or other neurodegenerative disorders.

DETAILED DESCRIPTION:
The goal of this study is to verify the effectiveness of the intensive-individual cognitive participation intervention (SCI-i) on the general cognitive functioning and specific cognitive functions of patients with mild or moderate cognitive decline affected by Alzheimer's dementia, Parkinson's and Multiple Sclerosis.

Participants will be subjected to cognitive training (tasks on attention, memory, language, executive functions, and visual-spatial functions) through software. They will take place using virtual cameras and virtual reality (VR) viewers. All subjects will undergo follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Alzheimer Disease, Multiple Sclerosis, Parkinson Disease
* Severity of mild to moderate cognitive impairment
* Sign informed consent

Exclusion Criteria:

* Important comorbidities with psychiatric syndromes
* Failure to sign the informed consent
* Atypical parkinsonisms
* Clinical conditions that involve vision-related problems.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Montreal cognitive assessment (MoCA) | up to 6 weeks
  MoCA (Montreal Cognitive Assessment or The MoCA Test) was validated as a highly sensitive tool for early detection of mild cognitive impairment (MCI) It quickly and accurately assesses: Short term memory; Visuospatial abilities; Executive functions; Attention, concentration, and working memory; Language; Orientation to time and place
  Results :
  26-30 points: No cognitive impairment 18-25 points: Mild cognitive impairment. 10-17 points: Moderate cognitive impairment. Fewer than 10 points: Severe cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Corallo, PSY, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Sicily, Italy